CLINICAL TRIAL: NCT01489254
Title: Multi-centre, Randomized, Double-blind, Placebo-controlled, Parallel-group, 9 Month, Equivalence Trial Comparing the Efficacy and Safety and Tolerability of GTR (Synthon BV) to Copaxone® (Teva) in Subjects With Relapsing Remitting Multiple Sclerosis Followed by an Open-label 15 Month GTR Treatment Part Evaluating the Long-term GTR Treatment Effects
Brief Title: Efficacy and Safety of GTR in Comparison to Copaxone®
Acronym: GATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Synthon BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GTR001; 2011-000888-27 (EudraCT Number)
Record Dates: First submitted 2011-12-08; First posted 2011-12-09 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis,; Relapsing-Remitting Multiple Sclerosis,; glatiramer acetate,; MRI,; lesions,; MS relapse rate,; Copaxone
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting | interventions — Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- GTR (Experimental): Drug
  Interventions: Drug: Glatiramer Acetate (GTR)
- Copaxone® (Active Comparator): Drug
  Interventions: Drug: Glatiramer Acetate (Copaxone®)
- Placebo (Placebo Comparator): Drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Glatiramer Acetate (GTR) — Glatiramer Acetate (GTR) 20 mg daily, for 9 months (Part 1) followed by additional 15 month treatment period (Part 2)
  Arms: GTR
Drug: Glatiramer Acetate (Copaxone®) — Glatiramer Acetate (Copaxone), 20 mg daily, for 9 months followed by additional 15 month GTR 20 mg daily treatment period (Part 2)
  Arms: Copaxone®
Drug: Placebo — Placebo (daily) for 9 months followed by additional 15 month GTR 20 mg daily treatment period (Part 2)
  Arms: Placebo

SUMMARY:
The purpose of this study is demonstrate that efficacy and safety of Synthon's glatiramer acetate (GTR) is equivalent to Copaxone® (Teva) in patients with relapsing remitting multiple sclerosis

DETAILED DESCRIPTION:
GTR is being developed by Synthon as a similar version of Copaxone®. GTR has a similar quantitative and qualitative composition as Copaxone®, with regard to active substance and excipients and is presented in the same dosage form (pre-filled syringe containing a solution for injection). Introduction of GTR is anticipated to have a price lowering effect and will give doctors and patients more choice in the pharmaceutical armamentarium for MS.

This trial consists of two parts:

Part 1 is a multi-country, multi-centre, randomized, double-blind, active and placebo-controlled, equivalence trial comparing the efficacy and safety and tolerability of GTR versus Copaxone® in subjects with RRMS. Eligible subjects will be randomly assigned to receive daily 20 mg GTR (Synthon BV), 20 mg Copaxone® (TEVA) or placebo for a period of 9 months.

In Part 2, the trial continues as an open-label uncontrolled trial to evaluate efficacy and safety of long-term treatment with GTR. Subjects completing the 9-month double-blind period will be treated with open-label 20 mg daily GTR for another 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign written Informed Consent;
* Female and male subjects aged 18-55 years inclusive at the time of Informed Consent signing;
* Diagnosis of RRMS according to the revised McDonald criteria;
* Expanded Disability Status Scale (EDSS) score of 0.0 up to and including 5.5;
* Neurologically stable with no evidence of relapse within 30 days prior to randomization;
* Experienced at least 1 relapse in the year before first screening assessment;
* At least 1 T1-weighted Gadolinium enhancing (T1-GdE) lesion on routine brain MRI taken within 3 months of starting screening or on screening brain MRI (as confirmed by central imaging laboratory;
* Having a routine brain MRI showing maximally 15 T1-GdE lesions if scan is taken without subject receiving immuno-modulatory treatment, or a routine brain MRI showing maximally 5 T1-GdE lesions when taken while on immuno-modulatory treatment, or a screening MRI showing maximally 15 T1-GdE lesions;
* Must decline initiation or continuation of treatment with other available disease-modifying drugs for MS, for whatever reason, after having been informed about their respective benefits and possible adverse events by the investigator;
* Female subjects of childbearing potential must agree to practice appropriate contraceptive methods as assessed by the investigator.

Exclusion Criteria:

* Any life-threatening, medically unstable or otherwise clinically significant condition or findings other than MS, in particular neoplastic disease, seizure disorders, or psychiatric disease;
* Any clinically significant deviation from reference ranges in laboratory tests;
* Positive laboratory test results for human immunodeficiency virus (HIV), HBsAg or HCV at screening;
* Any significant deviation from reference ranges for hepatic function;
* Positive urine drug screen or history of substance abuse within the year before screening (any use of illicit or prescription drugs or alcohol constituting an abuse pattern in the opinion of the investigator);
* Having been treated with or having received

  1. at any time:

     * glatiramer acetate, cladribine, rituximab, cyclophosphamide, alemtuzumab, or other immunosuppressive treatments with effects potentially lasting for more than 6 months
     * total lymphoid irradiation or bone marrow transplantation
  2. within one year before screening:

     * mitoxantrone, but subject cannot be enrolled when mitoxantrone was taken at a cumulative lifetime dosing above 100 mg/m2
  3. within 6 months before screening:

     * fingolimod, immunoglobulins and/or monoclonal antibodies (including natalizumab), leflunomide, or putative MS treatments
     * chronic oral or injected corticosteroids or injected ACTH (more than 30 consecutive days)
  4. within 3 months before screening:

     * azathioprine, methotrexate
     * plasma exchange
     * any other experimental intervention, in particular experimental drugs
  5. within 1 month before screening:

     * Interferon-β 1a or 1b
     * short-term oral or injectable corticosteroids for treatment of a relapse
     * short-term ACTH
* Having, in the opinion of the investigator, consecutively failed on efficacy grounds two full and adequate courses of accepted treatment modalities (normally at least one year of treatment for each);
* Pregnancy or breastfeeding;
* Known hypersensitivity to gadolinium-containing products, glatiramer acetate or mannitol;
* Having an estimated glomerular filtration rate (eGFR) < 50 mL/min/1.73m2;
* Inability to undergo (repeat) MRI investigations as judged by the investigator, e.g. due to claustrophobia, metal implants or fragments, tattoos or permanent make-up;
* Any reason why, in the investigator's opinion, the subject should not participate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 794 (Actual)
Dates: Start 2011-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (133):
- United States (7):
  - Synthon investigational site 112, Irvine, California
  - Synthon investigational site 120, Port Charlotte, Florida
  - Synthon investigational site 130, Sunrise, Florida
  - Synthon investigational site 107, Elk Grove Village, Illinois
  - Synthon investigational site 141, Raleigh, North Carolina
  - Synthon investigational site 106, Cleveland, Ohio
  - Synthon investigational site 135, Dayton, Ohio
- Belarus (7):
  - Synthon investigational site 401, Bitebsk
  - Synthon investigational site 403, Grodno
  - Synthon investigational site 402, Homyel
  - Synthon investigational site 404, Minsk
  - Synthon investigational site 407, Minsk
  - Synthon investigational site 408, Minsk
  - Synthon investigational site 405, Vitebsk
- Bosnia and Herzegovina (3):
  - Synthon investigational site 486, Banja Luka
  - Synthon investigational site 487, Sarajevo
  - Synthon investigational site 488, Tuzla
- Bulgaria (8):
  - Synthon investigational site 204, Pleven
  - Synthon investigational site 207, Pleven
  - Synthon investigational site 206, Plovdiv
  - Synthon investigational site 202, Sofia
  - Synthon investigational site 203, Sofia
  - Synthon investigational site 205, Sofia
  - Synthon investigational site 208, Sofia
  - Synthon investigational site 201, Varna
- Croatia (4):
  - Synthon investigational site 477, Osijek
  - Synthon investigational site 475, Zagreb
  - Synthon investigational site 476, Zagreb
  - Synthon investigational site 478, Zagreb
- Czechia (7):
  - Synthon investigational site 211, Brno
  - Synthon investigational site 217, Brno
  - Synthon investigational site 210, Olomouc
  - Synthon investigational site 212, Ostrava
  - Synthon investigational site 215, Prague
  - Synthon investigational site 216, Prague
  - Synthon investigational site 214, Teplice
- Estonia (2):
  - Synthon investigational site 297, Kohtla-Järve
  - Synthon investigational site 296, Tallinn
- Georgia (5):
  - Synthon investigational site 526, Tbilisi
  - Synthon investigational site 527, Tbilisi
  - Synthon investigational site 528, Tbilisi
  - Synthon investigational site 529, Tbilisi
  - Synthon investigational site 530, Tbilisi
- Synthon investigational site 227, Jena, Germany
- Italy (2):
  - Synthon investigational site 234, Coppito
  - Synthon investigational site 235, Naples
- Mexico (4):
  - Synthon investigational site 516, Guadalajara
  - Synthon investigational site 512, Mexico City
  - Synthon investigational site 514, Mexico City
  - Synthon investigational site 515, Morelia
- Moldova (4):
  - Synthon investigational site 547, Chisinau
  - Synthon investigational site 548, Chisinau
  - Synthon investigational site 549, Chisinau
  - Synthon investigational site 550, Chisinau
- Poland (12):
  - Synthon investigational site 244, Bialystok
  - Synthon investigational site 240, Katowice
  - Synthon investigational site 241, Katowice
  - Synthon investigational site 242, Katowice
  - Synthon investigational site 245, Katowice
  - Synthon investigational site 247, Lodz
  - Synthon investigational site 251, Lublin
  - Synthon investigational site 243, Olsztyn
  - Synthon investigational site 248, Poznan
  - Synthon investigational site 250, Szczecin
  - Synthon investigational site 246, Warsaw
  - Synthon investigational site 249, Wroclaw
- Romania (7):
  - Synthon investigational site 260, Bucharest
  - Synthon investigational site 262, Bucharest
  - Synthon investigational site 263, Bucharest
  - Synthon investigational site 264, Bucharest
  - Synthon investigational site 265, Bucharest
  - Synthon investigational site 266, Cluj-Napoca
  - Synthon investigational site 267, Timișoara
- Russia (26):
  - Synthon investigational site 438, Arkhangelsk
  - Synthon investigational site 435, Barnaul
  - Synthon investigational site 437, Belgorod
  - Synthon investigational site 445, Kaluga
  - Synthon investigational site 427, Kazan'
  - Synthon investigational site 432, Kemerovo
  - Synthon investigational site 447, Kirov
  - Synthon investigational site 446, Lipetsk
  - Synthon investigational site 571, Moscow
  - Synthon investigational site 428, Nizhny Novgorod
  - Synthon investigational site 429, Nizhny Novgorod
  - Synthon investigational site 434, Novosibirsk
  - Synthon investigational site 442, Novosibirsk
  - Synthon investigational site 444, Penza
  - Synthon investigational site 433, Pyatigorsk
  - Synthon investigational site 421, Saint Petersburg
  - Synthon investigational site 426, Saint Petersburg
  - Synthon investigational site 430, Saint Petersburg
  - Synthon investigational site 440, Saint Petersburg
  - Synthon investigational site 424, Samara
  - Synthon investigational site 420, Smolensk
  - Synthon investigational site 422, Tomsk
  - Synthon investigational site 441, Tver'
  - Synthon investigational site 425, Tyumen
  - Synthon investigational site 423, Ufa
  - Synthon investigational site 431, Yekaterinburg
- Serbia (4):
  - Synthon investigational site 450, Belgrade
  - Synthon investigational site 451, Belgrade
  - Synthon investigational site 453, Kragujevac
  - Synthon investigational site 452, Novi Sad
- South Africa (3):
  - Synthon investigational site 501, Cape Town
  - Synthon investigational site 505, Durban
  - Synthon investigational site 502, Pretoria
- Ukraine (23):
  - Synthon investigational site 474, Cherkassy
  - Synthon investigational site 459, Chernihiv
  - Synthon investigational site 463, Chernivtsi
  - Synthon investigational site 458, Dnipro
  - Synthon investigational site 472, Dnipro
  - Synthon investigational site 464, Donetsk
  - Synthon investigational site 468, Donetsk
  - Synthon investigational site 495, Ivano-Frankivsk
  - Synthon investigational site 461, Kharkiv
  - Synthon investigational site 469, Kharkiv
  - Synthon investigational site 455, Kyiv
  - Synthon investigational site 456, Kyiv
  - Synthon investigational site 496, Kyiv
  - Synthon investigational site 473, Lutsk
  - Synthon investigational site 462, Lviv
  - Synthon investigational site 466, Lviv
  - Synthon investigational site 497, Lviv
  - Synthon investigational site 498, Mariupol
  - Synthon investigational site 457, Odesa
  - Synthon investigational site 470, Poltava
  - Synthon investigational site 471, Uzhhorod
  - Synthon investigational site 465, Vinnytsia
  - Synthon investigational site 460, Zhytomyr
- United Kingdom (4):
  - Synthon investigational site 284, Sheffield
  - Synthon investigational site 281, Stoke-on-Trent
  - Synthon investigational site 283, Torquay
  - Synthon investigational site 280, Truro

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Cohen J, Belova A, Selmaj K, Wolf C, Sormani MP, Oberye J, van den Tweel E, Mulder R, Koper N, Voortman G, Barkhof F; Glatiramer Acetate Clinical Trial to Assess Equivalence With Copaxone (GATE) Study Group. Equivalence of Generic Glatiramer Acetate in Multiple Sclerosis: A Randomized Clinical Trial. JAMA Neurol. 2015 Dec;72(12):1433-41. doi: 10.1001/jamaneurol.2015.2154. PMID 26458034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomized at 118 investigational sites in 17 countries.
Pre-assignment Details: 1549 patients were assessed for eligibility of whom 796 subjects were randomized in a 4.3:4.3:1 ratio to receive generic glatiramer acetate (GTR), brand glatiramer acetate (Copaxone) or matching placebo. Two subjects were randomized to the generic glatiramer acetate group but did not start treatment and were not enrolled.
Groups:
- Glatiramer 20 mg: Glatiramer Acetate (GTR) 20 mg daily for 9 months
- Copaxone 20 mg: Glatiramer Acetate (Copaxone) 20 mg daily for 9 months
- Placebo: Placebo (daily) for 9 months
- Extension Glatiramer 20 mg: Glatiramer acetate (GTR) 20 mg daily for 15 months, open-label extension
Period: Double-blind Part
Arm/Group | Glatiramer 20 mg | Copaxone 20 mg | Placebo | Extension Glatiramer 20 mg
Started | 355 | 357 | 84 | 0
Completed | 330 | 324 | 81 | 0
Not Completed | 25 | 33 | 3 | 0
Not completed — Adverse Event | 7 | 2 | 2 | 0
Not completed — Pregnancy | 1 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 20 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — Other reasons for not completing study | 4 | 6 | 0 | 0
Period: Open-label Extension Part
Arm/Group | Glatiramer 20 mg | Copaxone 20 mg | Placebo | Extension Glatiramer 20 mg
Started | 0 | 0 | 0 | 728 (735 completed the DB part, 729 were eligible to continue in the OL part, 1 opted not to continue)
Completed | 0 | 0 | 0 | 670
Not Completed | 0 | 0 | 0 | 58
Not completed — Adverse Event | 0 | 0 | 0 | 10
Not completed — Pregnancy | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 30
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 9
Not completed — Other reasons for not completing study | 0 | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glatiramer 20 mg | Copaxone 20 mg | Placebo | Total
Number analyzed (Participants) | 353 | 357 | 84 | 794
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (8.6) | 33.8 (9.0) | 32.6 (8.7) | 33.1 (8.8)
Gender [Count of Participants; unit: Participants]
  Female | 233 | 238 | 57 | 528
  Male | 120 | 119 | 27 | 266
Time from first clinical event to randomization [Mean (Standard Deviation); unit: years] | 5.5 (5.3) | 6.4 (6.0) | 5.7 (6.0) | 5.9 (5.7)
Number of relapses in period within 2 year prior to signing ICF [Mean (Standard Deviation); unit: Number of relapses] | 1.9 (0.9) | 1.8 (0.9) | 1.9 (0.9) | 1.8 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: The Number of T1-Gadolinium Enhancing Lesions During Months 7-9
Description: The primary endpoint was the total number of gadolinium enhancing lesions (i.e., the cumulative number of new and persisting gadolinium enhancing lesions) during months 7 through 9.
Time Frame: 9 months
Population: Full Analyis Set (FAS): all randomized subjects who received at least 1 dose of trial medication
Measure: Mean (95% Confidence Interval); unit: Number of lesions
Arm/Group | Glatiramer 20 mg | Copaxone 20 mg | Placebo
Number analyzed (Participants) | 353 | 357 | 84
Number of lesions
  Sensitivity analysis - Number of Gd lesions | 0.42 [0.31 to 0.57] | 0.38 [0.28 to 0.52] | 0.82 [0.57 to 1.20]
  Equivalence analysis - Number of Gd lesions: number analyzed (Participants) | 353 | 357 | 0
  Equivalence analysis - Number of Gd lesions | 0.45 [0.34 to 0.59] | 0.41 [0.31 to 0.54] |
Statistical Analysis 1: Comparison: Glatiramer 20 mg vs Copaxone 20 mg vs Placebo; Estimates represent the mean total lesions during months 7 through 9 and were estimated from the fitted random effect generalized linear model (longitudinal model) with a negative binomial distribution and logaritmic link function. To assess study sensitivity, data of the active treatment groups and placebo were included in the model, resulting in the ratios and 95% CIs for the combined Glatiramer 20 mg and Copaxone 20 mg treatment group and the individual treatments over placebo; Test type: Non-Inferiority or Equivalence — To conclude study sensitivity the combined active treatment groups Glatiramer 20 mg and Copaxone 20 mg needed to be superior to placebo; Ratio (or Ratio of estimated means) = 0.488, 95% CI 2-sided [0.365 to 0.651] — Ratio of combined Glatiramer 20 mg + Copaxone 20 mg to placebo and 95% confidence interval
Statistical Analysis 2: Comparison: Glatiramer 20 mg vs Copaxone 20 mg; Estimates represent the mean total lesions during months 7 through 9 and were estimated from the fitted random effect generalized linear model (longitudinal model) with a negative binomial distribution and logaritmic link function including Glatiramer 20 mg and Copaxone 20 mg treatment groups to assess study equivalence; Test type: Non-Inferiority or Equivalence — To conclude equivalence between Glatiramer 20 mg and Copaxone 20 mg, efficacy in the combined active treatment groups needed to be superior to placebo (confirming study sensitivity) and the 2-sided 95% CI for the estimated ratio of Glatiramer 20 mg to Copaxone 20 mg needed to be fully enclosed in the prespecified equivalence margin (0.727 - 1.375); Ratio (or Ratio of estimated means) = 1.095, 95% CI 2-sided [0.883 to 1.360] — Ratio of Glatiramer 20 mg to Copaxone 20 mg and 95% confidence interval

ADVERSE EVENTS:
Time Frame: 9 months + 15 months
Description: The safety population consisted of all subjects who received at least 1 injection with study treatment.
Groups:
- Glatiramer 20 mg: Glatiramer Acetate (GTR) 20 mg daily for 9 months, double-blind
- Copaxone 20 mg: Glatiramer Acetate (Copaxone) 20 mg daily for 9 months, double-blind
- Placebo: Placebo (daily) for 9 months, double-blind
Arm/Group | Glatiramer 20 mg | Copaxone 20 mg | Placebo | Extension Glatiramer 20 mg
Serious Adverse Events (participants affected / at risk) | 12/353 | 17/357 | 2/84 | 22/728
Other Adverse Events (participants affected / at risk) | 110/353 | 121/357 | 29/84 | 90/728
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glatiramer 20 mg (N=353) | Copaxone 20 mg (N=357) | Placebo (N=84) | Extension Glatiramer 20 mg (N=728)
Anaphylactoid reaction (Immune system disorders) | 1 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 0 | 1 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Immediate post-injection reaction (General disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Abortion induced (Surgical and medical procedures) | 0 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Metastases to central nervous sytem (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Multiple sclerosis relapse (Nervous system disorders) | 2 | 4 | 0 | 5
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 1 | 0 | 0
Radiculitis cervical (Nervous system disorders) | 0 | 0 | 0 | 1
Secondary progressive multiple sclerosis (Nervous system disorders) | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Patellofemoral pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Glatiramer 20 mg (N=353) | Copaxone 20 mg (N=357) | Placebo (N=84) | Extension Glatiramer 20 mg (N=728)
Injection site reaction (General disorders) | 58 | 62 | 6 | 15
Immediate post-injection reaction (General disorders) | 24 | 17 | 0 | 11
Injection site swelling (General disorders) | 14 | 12 | 3 | 4
Injection site pain (General disorders) | 11 | 13 | 1 | 7
Injection site haematoma (General disorders) | 1 | 0 | 3 | 0
Injection site bruising (General disorders) | 0 | 0 | 3 | 1
Nasopharyngitis (Infections and infestations) | 13 | 23 | 6 | 39
Upper respiratory tract infection (Infections and infestations) | 6 | 6 | 3 | 5
Respiratory tract infection (Infections and infestations) | 2 | 4 | 4 | 4
Headache (Nervous system disorders) | 16 | 12 | 7 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Synthon's agreements with its investigators may vary. However, Synthon BV does not prohibit any investigator from publishing. Any publication from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.